CLINICAL TRIAL: NCT01227668
Title: Safety and Efficacy of Aripiprazole in the Long-term Maintenance Treatment of Pediatric Patients With Irritability Associated With Autistic Disorder
Brief Title: Phase IV Long-term Maintenance Study of Aripiprazole in the Treatment of Irritability Associated With Autistic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN138-603
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-03

CONDITIONS: Irritability Associated With Autistic Disorder
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 2-15 mg, once daily, 13-42 weeks
  Other Names: BMS-337039; Abilify
  Arms: Aripiprazole
Drug: Placebo — Tablets, Oral, 0 mg, once daily, 16 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether pediatric participants with irritability associated with autistic disorder who have responded to aripiprazole treatment will experience a relapse significantly later when continuing therapy with aripiprazole than will participants who receive placebo

DETAILED DESCRIPTION:
Phase 1: Single blind/ Phase 2: Double blind

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female children or adolescents, 6 to 17 years of age, inclusive, at the time of the baseline visit
* Meets current diagnostic criteria of the Diagnostic and Statistical Manual-of Mental Disorders IV-Text Revised for autistic disorder and displays behaviors such as tantrums, aggression, self-injurious behavior, or a combination of these problems. Diagnosis of autistic disorder will be confirmed by the Autism Diagnostic Interview-Revised.
* Participant or designated guardian or caregiver is able to comprehend and satisfactorily comply with the protocol requirements, in the opinion of the investigator.
* Demonstrates behaviors such as tantrums, aggression, or self-injury or a combination of these problems
* An Aberrant Behavior Checklist Irritability subscale score ≥18 AND a Clinical Global Impressions Severity score ≥4 at the Screening and Baseline Visits.
* Mental age of at least 24 months

Key Exclusion Criteria:

* Treatment resistant to neuroleptic medication, based on lack of therapeutic response to 2 different neuroleptics after treatment for at least 3 weeks each.
* Previous treatment with aripiprazole for at least 3 weeks duration at an adequate daily dose, without demonstrating a clinically meaningful response.
* Lifetime diagnosis of bipolar disorder, psychosis, or schizophrenia, or a current diagnosis of major depressive disorder
* Diagnosis of Pervasive Developmental Disorder-Not Otherwise Specified, Asperger's Syndrome, Rett's Syndrome, childhood disintegrative disorder, or Fragile X Syndrome
* History of neuroleptic malignant syndrome
* At significant risk for suicide based on history or routine psychiatric status examination
* A seizure within the past year
* History of severe head trauma or stroke
* History or current evidence of any unstable medical conditions that would expose the patient to undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial
* Weight lower than 15 kg
* Known allergy or hypersensitivity to aripiprazole or other dihidrocarbostyrils
* History of a clinically significant low white blood cell count or a drug-induced leukopenia/neutropenia
* Any other medically significant abnormal laboratory test or vital sign result or electrocardiogram finding

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- United States (38):
  - Harmonex Neuroscience Research, Inc, Dothan, Alabama
  - Southwest Autism Research And Resource Center, Phoenix, Arizona
  - Clinical Innovations, Inc., Costa Mesa, California
  - Behavioral Research Specialists, Llc, Glendale, California
  - Abbey Neuropsychology Clinic, Palo Alto, California
  - Ucsf - Lppi, San Francisco, California
  - Stanford University School Of Medicine, Stanford, California
  - Children'S National Medical Center, Washington D.C., District of Columbia
  - Sarkis Clinical Trials, Gainesville, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Florida Clinical Research Center, Llc, Maitland, Florida
  - Miami Children'S Hospital, Miami, Florida
  - University Of South Florida, Tampa, Florida
  - Institute For Behavioral Medicine, Llc, Smyrna, Georgia
  - Kootenai Behavioral Health Center, Coeur d'Alene, Idaho
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Lsu Health Sciences Center, Shreveport, Louisiana
  - Neurocare, Inc., Newton, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Center For Psychiatry And Behavioral Medicine, Inc, Las Vegas, Nevada
  - Clinical Research Center Of New Jersey, Gibbsboro, New Jersey
  - Children'S Specialized Hosp, Toms River, New Jersey
  - Stony Brook University School Of Medicine, Stony Brook, New York
  - Unc Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Nisonger Center, Columbus, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Ou Physician'S Child Study Center, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, Llc, Tulsa, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Drexel University College Of Medicine, Philadelphia, Pennsylvania
  - Western Psychiatric Institute And Clinic, Pittsburgh, Pennsylvania
  - Holston Medical Group, Kingsport, Tennessee
  - Insite Clinical Research, DeSoto, Texas
  - Ericksen Research And Development, Clinton, Utah
  - Childrens Specialty Gr., Pllc, Norfolk, Virginia
  - Virginia Treatment Center For Children, Richmond, Virginia

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Findling RL, Mankoski R, Timko K, Lears K, McCartney T, McQuade RD, Eudicone JM, Amatniek J, Marcus RN, Sheehan JJ. A randomized controlled trial investigating the safety and efficacy of aripiprazole in the long-term maintenance treatment of pediatric patients with irritability associated with autistic disorder. J Clin Psychiatry. 2014 Jan;75(1):22-30. doi: 10.4088/jcp.13m08500. PMID 24502859
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 215 participants enrolled, 58 discontinued during screening and before entry into Phase 1. Of the 58 who discontinued, 1 withdrew for an adverse event, 12 withdrew consent, 8 were lost to follow-up, 36 no longer met study criteria, and 1 withdrew for other reason.
Groups:
- Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose): Phase 1: Participants received an initial dose of aripiprazole 2 mg daily, titered up to 5, 10, or 15 mg once daily to optimize clinical benefit, for a maximum of 26 weeks.
  Phase 2: Aripiprazole was continued at the dose prescribed at the end of Phase 1, once daily for 16 weeks. The dose (within the range of 2-15 mg/day) could have been adjusted based on efficacy and tolerability.
- Placebo: Phase 2 only: Participants received placebo for 16 weeks.
Period: Phase 1 (Stabilization Phase)
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo
Started | 157 (Randomized) | 0
Received Treatment | 155 | 0
Completed | 85 | 0
Not Completed | 72 | 0
Not completed — Adverse Event | 12 | 0
Not completed — Withdrawal by Subject | 7 | 0
Not completed — Lost to Follow-up | 8 | 0
Not completed — Sponsor's administrative reason | 11 | 0
Not completed — No longer meets study criteria | 7 | 0
Not completed — Lack of Efficacy | 25 | 0
Not completed — Poor compliance/noncompliance | 2 | 0
Period: Phase 2 (Randomization Phase)
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo
Started | 41 (Randomized) | 44 (Randomized)
Received Treatment | 39 | 43
Completed | 22 | 19
Not Completed | 19 | 25
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 13 | 23
Not completed — Poor compliance/noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized to receive treatment in Phase 2
Groups:
- Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose): Phase 2: Aripiprazole was continued at the dose prescribed at the end of Phase 1, once daily for 16 weeks. The dose (within the range of 2-15 mg/day) could have been adjusted based on efficacy and tolerability.
- Placebo: Phase 2: Participants received placebo for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo | Total
Number analyzed (Participants) | 41 | 44 | 85
Age, Customized [Mean (Standard Deviation); unit: years] | 10.1 (2.80) | 10.8 (2.77) | 10.4 (2.79)
Age, Customized [Median (Full Range); unit: Years] | 10.0 [6 to 16] | 11.0 [6 to 17] | 10.0 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 30 | 38 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 31 | 28 | 59
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Relapsing by Week 16
Description: Time of relapse=date when patient meets relapse criteria. There are 4 definitions for relapse: 1. Patient meets the following criteria for 2 consecutive visits: (a) Aberrant Behavior Checklist Irritability score ≥25% than score at end of Phase 1 AND (b) Clinical Global Impression Improvement scale rating of 'Much Worse' or 'Very Much Worse' relative to rating at end of Phase 1. If relapse criteria met at 1 visit, 2nd visit should occur in about 1 week to reevaluate whether relapse criteria are still met. 2. Patient discontinues for "Lost to Follow-up" after a visit in which he or she met Definition 1 criteria (a&b). 3. Patient begins a prohibited drug (whether a study investigator or outside source prescribed) to treat worsening symptoms of irritability of autistic disorder after a visit where patient met Definition 1 criteria (a&b). 4. Patient discontinues due to hospitalization for worsening symptoms of irritability or due to lack of efficacy based on investigator's assessment.
Time Frame: From end of Phase 1 (Date of randomization) to Week 16 of Phase 2 and end of treatment
Population: All participants who were randomized in Phase 2
Measure: Number; unit: Percentage of participants
Groups:
- Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose): Phase 2: Participants continued aripiprazole at the dose prescribed at the end of Phase 1, once daily for 16 weeks. The dose (within the range of 2-15 mg/day) could have been adjusted based on efficacy and tolerability.
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo
Number analyzed (Participants) | 41 | 44
Percentage of participants | 32 (NA) [NA to NA] | 50 [42 to NA]
Statistical Analysis 1: Comparison: Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) vs Placebo; Test type: Superiority or Other; p = 0.097, Stratified log rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.28 to 1.12]

2. Secondary Outcome: Adjusted Mean Change From Baseline to Week 16 on the Aberrant Behavior Checklist Irritability (ABC-I) Subscale Score (Last Observation Carried Forward [LOCF])
Description: ABC is an informant-based checklist used to assess and classify problem behaviors of children and adolescents with mental retardation. The 58 items are rated on a 4-point scale (0=not at all a problem to 3=the problem is severe in degree), and resolve into 5 subscales: 1) irritability, agitation; 2) lethargy, social withdrawal; 3) stereotypic behavior; 4) hyperactivity, noncompliance; and 5) inappropriate speech. The ABC can be completed by parents, special educators, psychologists, direct caregivers, nurses, and others knowing the participant. Psychometric assessment of the ABC indicates that its subscales have high internal consistency, adequate reliability, and established validity. The ABC-I Subscale Score ranges from 0 to 45, with a negative change in score signifying improvement. LOCF data set includes data recorded at a given visit or, if no observation was recorded at that visit, data carried forward from the prior visit. chg=change; BL=baseline; APR=aripiprazole; vs=versus.
Time Frame: From Baseline (end of Phase 1) to Week 16 of Phase 2
Population: All participants who were randomized and took at least 1 dose of double-blind medication in Phase 2 and who had at least 1 efficacy evaluation after the start of Phase 2 study drug.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo
Number analyzed (Participants) | 39 | 43
Units on a scale | 5.2 (1.61) [0.0 to 10.0] | 9.6 (1.56) [1.0 to 19.0]
Statistical Analysis 1: Comparison: Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) vs Placebo; Test type: Superiority or Other; p = 0.051, ANCOVA — For secondary endpoints, hierarchical testing aimed to keep the overall experiment-wise type I error rate to <=0.05. Difference in chg from BL was tested at 0.05 significance only if APR arm significantly differed vs placebo from primary analysis; Mean Difference (Final Values) = -4.40, 95% CI 2-sided [-8.82 to 0.02]

3. Secondary Outcome: Change From Baseline in Mean Clinical Global Impression Improvement (CGI-I) Scale Score at Week 16 (Last Observation Carried Forward [LOCF])
Description: CG-I rating scale permits global evaluation of patient's improvement over time. At baseline (BL), CGI Severity of Illness assessment is performed, in which the clinician rates severity of patient's condition on a 7-point scale ranging from 1=no symptoms to 7=very severe symptoms. Higher total score=worse symptoms. At subsequent visits, clinician assesses patient's improvement relative to symptoms at baseline on CGI-I 7-point scale ranging from 1=very much improved to 7=very much worse. Since the drug targets irritability symptoms, the CGI focuses on severity of irritability secondary to autistic disorder. Lower score=more improved symptoms. LOCF data set includes data recorded at a given visit or, if nothing recorded, data areccarried forward from the prior visit. For secondary endpoints (endpt), hierarchical testing was used to keep overall experiment-wise type I error rate to <=0.05. diff=difference; IS=irritability scale; PA=primary analysis; signif=significance/significantly.
Time Frame: From Baseline (end of Phase 1) to Week 16 of Phase 2
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose): Phase 2: Participants continued aripiprazole (ARP) at the dose prescribed at the end of Phase 1, once daily for 16 weeks. The dose (within the range of 2-15 mg/day) could have been adjusted based on efficacy and tolerability.
- Placebo: Phase 2 only: Participants received placebo (pb)for 16 weeks.
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo
Number analyzed (Participants) | 39 | 43
Units on a scale | 4.2 (0.26) | 4.8 (0.26)
Statistical Analysis 1: Comparison: Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) vs Placebo; Test type: Superiority or Other; p = 0.090, ANCOVA — Treatment diff in chg from BL to endpnt in IS score was tested at 0.05 signif only if ARP arm signif differed vs pb from PA. Thus, if ARP arm signif differed vs pb in IS score, treatment diff in mean CGI-I score at endpnt was tested at 0.05 signfnce; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.3 to 0.1]

4. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), and Adverse Events (AEs) Leading to Discontinuation During Phase 1
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Weekly from Week 1 to Week 26 and continuously to end of treatment
Population: All participants who took at least 1 dose of single-blind aripiprazole in Phase 1
Measure: Number; unit: Participants
Groups:
- Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose): Phase 1: Participants received an initial dose of aripiprazole 2 mg daily, titered up to 5, 10, or 15 mg once daily to optimize clinical benefit, for a maximum of 26 weeks.
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose)
Number analyzed (Participants) | 155
Participants
  Death | 0
  SAEs | 1
  AEs leading to discontinuation | 13

5. Other Pre Specified Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Treatment-related AEs During Phase 2
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: Weekly from Weeks 1 through 16 (end of treatment) of Phase 2
Population: All participants who were randomized and took at least 1 dose of double-blind medication in Phase 2
Measure: Number; unit: Participants
Arm/Group | Aripiprazole, 2-15 mg Once Daily (Titered to Optimum Dose) | Placebo
Number analyzed (Participants) | 39 | 43
Participants
  Death | 0 | 0
  SAEs | 0 | 0
  AEs leading to discontinuation | 0 | 0
  Treatment-related AEs | 9 | 6

ADVERSE EVENTS:
Groups:
- Aripiprazole, 2-15 mg (Phase 1): Phase 1: Participants received an initial dose of aripiprazole 2 mg daily, titered up to 5, 10, or 15 mg once daily to optimize clinical benefit, for a maximum of 26 weeks.
- Aripiprazole, 2-15 mg (Phase 2): Phase 2: Participants continued aripiprazole at the dose prescribed at the end of Phase 1, once daily for 16 weeks. The dose (within the range of 2-15 mg/day) could have been adjusted based on efficacy and tolerability.
- Placebo (Phase 2 Only): Phase 2 only: Participants received placebo for 16 weeks.
Arm/Group | Aripiprazole, 2-15 mg (Phase 1) | Aripiprazole, 2-15 mg (Phase 2) | Placebo (Phase 2 Only)
Serious Adverse Events (participants affected / at risk) | 1/155 | 0/39 | 0/43
Other Adverse Events (participants affected / at risk) | 112/155 | 11/39 | 5/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole, 2-15 mg (Phase 1) (N=155) | Aripiprazole, 2-15 mg (Phase 2) (N=39) | Placebo (Phase 2 Only) (N=43)
Aggression (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole, 2-15 mg (Phase 1) (N=155) | Aripiprazole, 2-15 mg (Phase 2) (N=39) | Placebo (Phase 2 Only) (N=43)
Fatigue (General disorders) | 13 | 1 | 0
Tremor (Nervous system disorders) | 10 | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 2 | 0
Movement disorder (Nervous system disorders) | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 22 | 2 | 2
Insomnia (Psychiatric disorders) | 13 | 1 | 1
Pyrexia (General disorders) | 8 | 1 | 0
Somnolence (Nervous system disorders) | 23 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 20 | 1 | 2
Lethargy (Nervous system disorders) | 8 | 0 | 0
Aggression (Psychiatric disorders) | 8 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 1 | 0
Headache (Nervous system disorders) | 8 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 16 | 4 | 1
Weight increased (Investigations) | 39 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.